CLINICAL TRIAL: NCT07327450
Title: Coaching Doctors and Nurses to Improve Ethical Decision-making in Team: a Stepped Wedge Cluster Randomized Trial in 10 Departments of the Ghent University Hospital.
Brief Title: Coaching Doctors and Nurses to Improve Ethical Decision-making in Team
Acronym: CODE II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: ONZ-2025-0602
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Decision Making ,Shared; Leadership; End of Life Communication; End of Life Decision Making; End of Life Patients; Ethical Sensitivities; Coaching
Keywords: Coaching; Shared decision-making; Goal-oriented care; Ethical climate; Leaderschip; Communication; End-of-life
MeSH Terms: conditions — Communication; Death

STUDY DESIGN:
Intervention Model Description: In total 50 to 75 junior doctors, 50 to 75 senior doctors (including medical head of department), 300 to 500 nurses (including head nurses) and 100 to 200 allied health professionals working in 10 departments of the Ghent University Hospital are eligible for this study and about 350 to 700 adult patients potentially receiving excessive treatment who did not yet receive a written DNI-DNACPR order together with one of their relatives. Stepped wedge cluster randomized trial in 10 hospital wards combined with pre- and post-measurement of the ethical climate.
Who Masked: Participant
Masking Description: Patients will be blinded to the 4 months intervention period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator)
  Interventions: Other: Usual Care Group
- CODE II intervention (Experimental)
  Interventions: Behavioral: CODE II intervention

INTERVENTIONS:
Other: Usual Care Group — The control group will receive usual care in which the quality of the ethical decision-making is determined by the clinical team according to their usual pratice. Except from a treatment-limitation-decisions guideline which focuses on the legal and deontological framework, no other guideline with regard to ethical decision-making has been implemented at the Ghent University Hospital.
  Arms: Usual care
Behavioral: CODE II intervention — 1) One interactive session of two hours focusing on the concepts of medical-ethical decision-making, the psychological challenge of dealing with ethically sensitive medical topics, empowering leadership and the importance of "speaking up" within the team. 2) Every clinician will be invited to provide perceptions of excessive treatment via the electronic patient file. Once a patient is identified by two or more different clinicians, an email will be sent to coaches and the clinicians in charge of the PET during intervention period. 3) The 4 months coaching intervention will consist of : a. Doctors and head nurses : individual coaching sessions in self-reflective and empowering leadership and in managing groups dynamics with regard to ethical decision-making in team about PET patients. b. All clinicians : multidisciplinary coaching during work shift hand-overs and structured metareflective sessions on specific themes related to ethical decision-making in team about PET.
  Arms: CODE II intervention

SUMMARY:
Literature and a pilot study performed in 2019 indicate room for enhancing openness to discuss ethical sensitive issues within and between teams, and improving goal-oriented care and decision-making for the benefit of the patient at end-of-life, worldwide and more specifically in Belgium and in the Ghent University Hospital. The CODE study intervention performed in 2021 suggests already an improvement in goal oriented care operationalized via written Do-Not-Intubate and Do-Not-Attempt Cardio-Pulmonary Resuscitation (DNI-DNACPR orders in our hospital. In this study, we found a nearly doubling of the incidence in written DNI-DNACPR in patient potentially receiving excessive treatment (PET) (from 19.7% to 29.7%, p<0.001) and in patients hospitalized for the first time (from 1.9% to 3.4%, p=0.011) without increasing one-year mortality, after coaching doctors during 4 months in self-reflective and empowering leadership, and coping with group dynamics. However, we found no improvement in the perception of the quality of the ethical climate by clinicians, more specifically by nurses. Despite the fact that ethical decision-making is considered a strategic priority in the Ghent University Hospital and an intense communication campaign, clinicians identified also a much smaller number of PET during this interventional study than during our observational pilot study in 2019. Although fading attention for the study over time and visibility of the electronic CODE alert to identify PET was claimed as the main reasons by 75% and 50.7% of the nurses, respectively, 95% expressed the desire to keep on using this alert in the future. This underscores a deeper concern in nurses. More than 40% expressed fear of blaming doctors or skepticism regarding the impact of identifying PET. Nonetheless, 35% acknowledged improvement in interdisciplinary meetings about end-of-life issues since study initiation. These findings highlights the need to additionally coach the entire team in future studies. Indeed, creating a safe climate which enhances inter-professional shared decision-making for the benefit of the patient requires both, specific self-reflective and empowering leadership skills in doctors and head nurses (including the management of group dynamics in the interdisciplinary team), and confidence in speaking up in nurses and other health care professionals. This is what we want to develop with this intervention. These skills will also help clinicians during patient and family meetings which will enable clinicians to better take into account the patient's and family's wishes.

DETAILED DESCRIPTION:
See protocol

ELIGIBILITY:
Inclusion Criteria:

* Patients potentially receiving excessive treatment (PET) who are identified by clinicians during their first hospitalization. PET is defined as a patient in whom 2 or more clinicians doubt whether the treatment or treatment limitation code is consistent with their expected survival or quality of life (= "too much" or "excessive treatment") or whether the treatment limitation code is in line with the patient's or relatives' goals.
* Family members of PET
* Junior and senior doctors (including Department Heads) taking care of hospitalized patients
* Nurses (including head nurses) taking care of hospitalized patients
* Allied health professionals (psychologists, physical therapists, speech therapists, occupational therapists, social workers, spiritual care providers) taking care of hospitalized patients
* PET admitted / clinicians working in the 10 participating departments of of the Ghent University Hospital (Cardiology, Gastro-enterology and Hepatology, General Internal Medicine, Geriatrics, Hematology, Medical Oncology, Neurology, Nephrology (including dialysis unit), Pulmonology and the Medical ICU)

Exclusion Criteria:

* PET with a previous written DNI-DNACPR order
* Patients and family members of PET who are less than 18 years old and persons who cannot understand Ducth questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of written DNI-DNACPR order between hospital admission and the end of the first hospital stay | At the end of the 12 months study period
  Patient-specific endpoint
Ethical decision-making climate questionnaire (EDMCQ) | at the start and the end of the 12 month study period
  Clinician specific endpoint. Factorscores on 7 domains, which is normally distributed, centred at mean of zero, with standard deviation 5.5 (minimum score -25, maximum score 25). Higher scores indicate higher quality of interdisciplinary ethical decision-making

SECONDARY OUTCOMES:
Hospital Consumer Assessment of Healthcare Providers and Systems instrument | 3 weeks after the patient's hospital discharge
  Patient-specific endpoint. Patients rate the quality of their hospital stay on a scale of 0 (worst) to 10 (best) and indicate whether they would recommend their hospital to family and friends.
Sinclair Compassion Questionnaire-Short Form (SCQ-SF) | 3 weeks after the patient's hospital discharge
  Patient-specific endpoint. The SCQ is a validated instrument for quantifying compassion in healthcare from multiple perspectives (e.g., patients, family, clinicians). It studies outcomes valued by the patient such as 'feeling heard and understood by their clinician' and 'being valued as a person'. The Belgian version of the 5-item SCQ-SF (Sinclair Compassion Questionnaire-Short Form) is used with each item rating on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score is calculated as the mean of the five items, resulting in a theoretical range from 1 to 5. A higher SCQ score is indicative of higher compassionate care.
Satisfaction according to the European Family Satisfaction in the ICU (Euro-FS) score | 3 weeks after the patient's hospital discharge
  Patient-specific endpoint. Validated 18 item questionnaire covering satisfaction with 4 domains: communication, empathy, symptom management and decision-making. The investigators will use the single-item assessment of satisfaction of this score raning from 0 to 10. higher values indicate higher satisfaction.
Hospital Anxiety and Depression Scale (HADS) | 3 weeks after hospital discharge
  Patient-specific endpoint. Validated 14-item self-report assessment with subscales for anxiety and depression. Each domain has a score range of 0-21 with the following interpretation: 0-7 normal, 8-10 mild, 11-21 moderate to severe
European quality of dying and death family questionnaire (Euro-QODD) | 3 weeks after the patient's hospital discharge
  Patient-specific endpoint filled out by the relatives. Euro-QDDD family is a 14 item questionnaire to allow relatives to assess patients quality of dying and death.
Pain according to the Numeral Rating scale (NRS) : sum of the average daily score up to the end of the first hospital stay | at the end of the 12 month study period
  Patient-specific endpoint; Single-item assessment of pain ranging from 0 (no pain) to 10 (worst possible pain)
Pain according to the Numeral Rating Scale (NRS) : number of days with an average score > 3 up to the end of the first hospital stay | at the end of the 12 month study period
  Patient-specific endpoint. Single-item assessment of pain raging from 0 (no pain) to 10 (worst possible pain).
Incidence of death up to one year after first hospital admission | 12 months after first hospital admission
  Patient-specific endpoint
Percentage of patients who achieved the combined one year outcome (dead, not at home or utility <0.5 according to the European Quality-of-life 5 dimension instrument(Euro-QOL-5D)) | 12 months after first hospital admission
  Patient-specific endpoint. Euro-QOL-5D measures health-related quality of life, with possibility of conversion of each health state in a utility index (range -0.1584 to 1.000). This questionnaire measures health in five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
Potentially inappropriate or burdensome treatments : incidence of achieving the combined patient burdensome treatments outcome (achieving outcome 13,14,15,16,17,18 or 19) up to one year after the first hospitalisation | At the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdensome treatments : incidence of receiving cardio-pulmonary resuscitation up to one year after the first hospitalisation | at the end of the 12 months study period
  Patient-specific endpoint
Potentially inappropriate or burdensome treatments : incidence of admission in the intensive care unit up to one year after the first hospitalisation | At the end of the 12 month study period
  Patient-specific endpoint
Potentially inappropriate or burdensome treatments : incidence of receiving invasive mechanical ventilation up to one year after the first hospitalisation | At the end of the 12 month study period
  Patient-specific endpoint
Potentially inappropriate or burdensome treatments : incidence of receiving dialysis up to one year after the first hospitalisation | At the end of the 12 month study period
  Patient-specific endpoint
Potentially inappropriate or burdensome treatments : incidence of receiving a surgical procedure up to one year after the first hospitalisation | At the end of the 12 month study period
  Patient-specific endpoint
Potentially inappropriate or burdensome treatments : incidence of receiving chemotherapy up to one year after the first hospitalisation | At the end of the 12 month study period
  Patient-specific endpoint
Potentially inappropriate or burdensome treatments : incidence of receiving radiotherapy up to one year after the first hospitalisation | At the end of the 12 months study period
  Patient-specific endpoint
Hospital Consumer Assessment of Healthcare Providers and Systems instrument | 3 weeks after the patient's hospital discharge
  Family-specific endpoint. Family rate the quality of their hospital stay on a scale of 0 (worst) to 10 (best) and indicate whether they would recommend their hospital to family and friends.
Sinclair Compassion Questionnaire-Short Form (SCQ-SF) | 3 weeks after the patient's hospital discharge
  Family-specific endpoint. The SCQ is a validated instrument for quantifying compassion in healthcare from multiple perspectives (e.g., patients, family, clinicians). It studies outcomes valued by the patient such as "feeling heard and understood by their clinicians" and "being valued as a person". The Belgian version of the 5-item SCQ-SF (Sinclair Compassion Questionnaire-Short Form) is used with each item rating on a five-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The total score is calculated as the mean of the five items, resulting in a theoretical range from 1 to 5. A higher SCQ score is indicative of higher compassionate care.
Satisfaction according to the European Family Satisfaction in the ICU (Euro-FS) score | 3 weeks after the patient's hospital discharge
  Family-specific endpoint. Validated 18 item questionnaire covering satisfaction with 4 domains: communication, empathy, symptom management and decision-making. The investigators will use the single-item assessment of satisfaction of this score raning from 0 to 10. higher values indicate higher satisfaction.
Hospital Anxiety and Depression Scale (HADS) | 3 weeks after the patient's hospital discharge
  Family-specific endpoint. Validated 14-item self-report assessment with subscales for anxiety and depression. Each domain has a score range of 0-21 with the following interpretation: 0-7 normal, 8-10 mild, 11-21 moderate to severe
Differences in EDMCQ between doctors and nurses | at the start and end of the 12 month study period
  Clinician spefic endpoint. Factorscores on 7 domains, which is normally distributed, centred at mean zero, with standard deviation 5.5 (minimum score -25, maximum score 25). Higher difference in scores between doctors and nurses indicate a greater gap in the perception of the ethical climate between roles.
Percentage of (mild-moderate-severe-extreme) stress related to a perception of excessive treatment | At the end of the 12 month study period
  Clinician-specific endpoint
Percentage of clinicians with intention of leaving their job | At the start and end of the 12 month study period
  Clinician-specific endpoint
Percentage of clinicians with sick leave | At the start and end of the 12 month study period
  Team-specific endpoint
Ethical pratice score | At the start and end of the 12 month study period
  Team-specific endpoint. This score consists of 12 items. The investigators will use the 10 department specific items (minus the 2 country-specific items). This score ranges between 0 to 10 with higher scores indicating a higher degree of ethical pratice organization
Incidence of written DNI-DNACPR order between hospital admission and the end of the first hospital stay in the overall patient population admitted in the participating wards | At the end of the 12 months study period
  Patient-specific endpoint
Incidence of death up to one year after first hospital admission in the overall patient population admitted in the participating wards | At the end of the 12 month study period
  Patient-specific endpoint
Health-care utilization : total number of chemotherapeutic treatments up to one year after the first hospital admission | 12 months after the first hospital admission
  Society-specific endpoint

OTHER OUTCOMES:
Health-care utilization : total hospital cost by the hospital billing record up to one year after the first hospital admission | 12 months after first hospital admission
  Society-level endpoint
Health-care utilization : total number of emergency department visits up to one year after the first hospital admission | 12 months after first hospital admission
  Society-specific endpoint
Health-care utilization : total number of hospitalizations up to one year after the first hospital admission | 12 months after first hospital admission
  Society-specific endpoint
Health-care utilization : total number of admission in the Intensive care Unit up to one year after the first hospital admission | 12 months after first hospital admission
  Society-specific endpoint
Health-care utilization : total number of days in the hospital up to one year after the first hospital admission | 12 months after first hospital admission
  Society-specific endpoint
Health-care utilization : total number of dialysis sessions up to one year after the first hospital admission | 12 months after the fisrt hospital admission
  Society-specific endpoint
Health-care utilization : total number of surgical procedures up to one year after the first hospital admission | 12 months after the first hospital admission
  Society-specific endpoint
Health-care utilization : total number of radiotherapeutic sessions up to one year after the first hospital admission | 12 months after the first hospital admission
  Society-specific endpoint
Health-care utilization : total number of radiologic investigations up to one year after the first hospital admission | 12 months after the first hospital admissions
  Society-specific endpoint
Health-care utilization : total number of blood analyses up to one year after the first hospital admission | 12 months after the first hospital admission
  Society-specific endpoint
Health-care utilization : total number of chemotherapeutic treatments up to one year after the first hospital admission | 12 months after the first hospital admission
  Society-specific endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No
In order to guaranty the entire safety of the participating departments and as such the change management trajectories of these departments, IPD will not be shared. Specific departments admit specific patient population : therefore, the quality of the ethical climate per department cannot be anonymized.

REFERENCES:
- [Background] Gerritsen RT, Koopmans M, Hofhuis JG, Curtis JR, Jensen HI, Zijlstra JG, Engelberg RA, Spronk PE. Comparing Quality of Dying and Death Perceived by Family Members and Nurses for Patients Dying in US and Dutch ICUs. Chest. 2017 Feb;151(2):298-307. doi: 10.1016/j.chest.2016.09.003. Epub 2016 Sep 19. PMID 27660153
- [Background] Spinhoven P, Ormel J, Sloekers PP, Kempen GI, Speckens AE, Van Hemert AM. A validation study of the Hospital Anxiety and Depression Scale (HADS) in different groups of Dutch subjects. Psychol Med. 1997 Mar;27(2):363-70. doi: 10.1017/s0033291796004382. PMID 9089829
- [Background] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Background] Jensen HI, Gerritsen RT, Koopmans M, Downey L, Engelberg RA, Curtis JR, Spronk PE, Zijlstra JG, Ording H. Satisfaction with quality of ICU care for patients and families: the euroQ2 project. Crit Care. 2017 Sep 7;21(1):239. doi: 10.1186/s13054-017-1826-7. PMID 28882192
- [Background] Sinclair S, Kondejewski J, Hack TF, Boss HCD, MacInnis CC. What is the Most Valid and Reliable Compassion Measure in Healthcare? An Updated Comprehensive and Critical Review. Patient. 2022 Jul;15(4):399-421. doi: 10.1007/s40271-022-00571-1. Epub 2022 Feb 2. PMID 35107822
- [Background] US Department of Health and Human Services. Hospital compare quality of care. 2011. www.hospitalcompare.hhs.gov
- [Background] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Background] Benoit DD, De Pauw A, Jacobs C, Moors I, Offner F, Velghe A, Van Den Noortgate N, Depuydt P, Druwe P, Hemelsoet D, Meurs A, Malotaux J, Van Biesen W, Verbeke F, Derom E, Stevens D, De Pauw M, Tromp F, Van Vlierberghe H, Callebout E, Goethals K, Lievrouw A, Liu L, Manesse F, Vanheule S, Piers R. Coaching doctors to improve ethical decision-making in adult hospitalized patients potentially receiving excessive treatment. The CODE stepped-wedge cluster randomized controlled trial. Intensive Care Med. 2024 Oct;50(10):1635-1646. doi: 10.1007/s00134-024-07588-0. Epub 2024 Sep 4. PMID 39230678
- [Background] Benoit DD, Vanheule S, Manesse F, Anseel F, De Soete G, Goethals K, Lievrouw A, Vansteelandt S, De Haan E, Piers R; CODE study group. Coaching doctors to improve ethical decision-making in adult hospitalised patients potentially receiving excessive treatment: Study protocol for a stepped wedge cluster randomised controlled trial. PLoS One. 2023 Mar 21;18(3):e0281447. doi: 10.1371/journal.pone.0281447. eCollection 2023. PMID 36943825
- [Background] Benoit DD, Jensen HI, Malmgren J, Metaxa V, Reyners AK, Darmon M, Rusinova K, Talmor D, Meert AP, Cancelliere L, Zubek L, Maia P, Michalsen A, Vanheule S, Kompanje EJO, Decruyenaere J, Vandenberghe S, Vansteelandt S, Gadeyne B, Van den Bulcke B, Azoulay E, Piers RD; DISPROPRICUS study group of the Ethics Section of the European Society of Intensive Care Medicine. Outcome in patients perceived as receiving excessive care across different ethical climates: a prospective study in 68 intensive care units in Europe and the USA. Intensive Care Med. 2018 Jul;44(7):1039-1049. doi: 10.1007/s00134-018-5231-8. Epub 2018 May 28. PMID 29808345
- [Background] Bekelman JE, Halpern SD, Blankart CR, Bynum JP, Cohen J, Fowler R, Kaasa S, Kwietniewski L, Melberg HO, Onwuteaka-Philipsen B, Oosterveld-Vlug M, Pring A, Schreyogg J, Ulrich CM, Verne J, Wunsch H, Emanuel EJ; International Consortium for End-of-Life Research (ICELR). Comparison of Site of Death, Health Care Utilization, and Hospital Expenditures for Patients Dying With Cancer in 7 Developed Countries. JAMA. 2016 Jan 19;315(3):272-83. doi: 10.1001/jama.2015.18603. PMID 26784775
- [Background] Kompanje EJ, Piers RD, Benoit DD. Causes and consequences of disproportionate care in intensive care medicine. Curr Opin Crit Care. 2013 Dec;19(6):630-5. doi: 10.1097/MCC.0000000000000026. PMID 24240830
- [Background] Curtis JR, Vincent JL. Ethics and end-of-life care for adults in the intensive care unit. Lancet. 2010 Oct 16;376(9749):1347-53. doi: 10.1016/S0140-6736(10)60143-2. Epub 2010 Oct 11. PMID 20934213